CLINICAL TRIAL: NCT06946290
Title: Intertransverse Process Block to Improve Quality of Recovery and Pain Management in Adult Cardiac Surgical Patients: a Prospective Double-Blinded Randomized Controlled Trial
Brief Title: Intertransverse Process Block to Improve Quality of Recovery and Pain Management in Adult Cardiac Surgical Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, WONG MAN KIN, Consultant Anaesthesiologist, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITPB - chronic pain
Record Dates: First submitted 2025-03-25; First posted 2025-04-27 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Chronic Postsurgical Pain
Keywords: ITPB; Intertransverse process block; Chronic postsurgical pain; Cardiac surgery; quality of recovery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ITPB group (Experimental): Intertransverse process block is performed on patients with injection of 20ml 0.25% levobupivacaine at the retro-SCTL space after a test bolus of 1-2ml 0.9% normal saline. The same procedure is repeated on the other side with same volume of study medication.
  Interventions: Procedure: Intertransverse process block
- Sham block group (Sham Comparator): Sham intertransverse process block is performed on patients with injection of 20ml placebo at the retro-SCTL space after a test bolus of 1-2ml 0.9% normal saline. The same procedure is repeated on the other side with same volume of study medication.
  Interventions: Procedure: Sham block

INTERVENTIONS:
Procedure: Intertransverse process block — All blocks are performed by an anaesthesiologist who had previously performed ≥50 successful ITPB blocks, using Philips EPIQ ultrasound system, with a curved array transducer (C5-1), and 80mm echogenic nerve block needle. ITPB is performed with the patients positioned in a lateral decubitus position. The target intervertebral level (T4-5) is identified and marked in the preview ultrasound scan. The transducer is placed 2-3 cm lateral to the spinous process. Under strict asepsis, a single-level (T4-5) ultrasound-guided ITPB is performed with the in-plane insertion of the block needle from lateral to medial direction until its tip is at the medial aspect of the retro-SCTL space. After confirming the needle position by distension of the retro-SCTL space after a test bolus injection of 1-2 ml 0.9% normal saline, 20 ml 0.25% levobupivacaine is injected via the nerve block needle in small aliquots. The same procedure is repeated on the other side with the same volume of study medication.
  Arms: ITPB group
Procedure: Sham block — All blocks are performed by an anaesthesiologist who had previously performed ≥50 successful ITPB blocks, using Philips EPIQ ultrasound system, with a curved array transducer (C5-1), and 80mm echogenic nerve block needle (SonoTAP; PAJUNK, Germany). ITPB is performed with the patients positioned in a lateral decubitus position. The target intervertebral level (T4-5) is identified and marked in the preview ultrasound scan. The transducer is placed 2-3 cm lateral to the spinous process. Under strict asepsis, a single-level (T4-5) ultrasound-guided ITPB is performed with the in-plane insertion of the block needle from lateral to medial direction until its tip is at the medial aspect of the retro-SCTL space. After confirming the needle position by distension of the retro-SCTL space after a test bolus injection of 1-2 ml 0.9% normal saline, 20 ml placebo is injected via the nerve block needle in small aliquots. The same procedure is repeated on the other side with the same volume study drug.
  Arms: Sham block group

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of intertransverse process block (ITPB) in improving quality of recovery and potentially preventing chronic postsurgical pain (CPSP) in adult patients undergoing elective cardiac surgery (e.g., coronary artery bypass graft [CABG], valve repair/replacement, or combined CABG/valve procedures).

The main questions it aims to answer are:

1. To investigate the quality of recovery after cardiac surgery, and its analgesic efficacy in the immediate postoperative period
2. To investigate the efficacy of intertransverse process block (ITPB) on CPSP after cardiac surgery by determining the incidence of CPSP at 3 month, defined as persistent pain that was not present before surgery or that had different characteristics, and other possible causes of pain are excluded.
3. To investigate the efficacy of ITPB on the incidence of CPSP at 6 month, 12 month, and the pain interference (sensory and affective components, physical activities) at 3 month, 6 month and 12 month after surgery

DETAILED DESCRIPTION:
Introduction:

The cornerstone of modern pain management in cardiac surgery lies in proactively preventing the development of chronic postsurgical pain (CPSP). This paradigm shift emphasizes pre-emptive interventions to disrupt the cascade of events and central sensitization that transform acute postoperative pain into a persistent, debilitating condition. CPSP, a significant and often underestimated consequence of cardiac surgery, affects a substantial proportion of patients, with prevalence rates ranging from 28% to 56% in the years following surgery. Its impact extends beyond mere discomfort, significantly impairing daily function, reducing quality of life, and imposing a substantial economic burden on the healthcare system.

The pathophysiology of CPSP involves a complex interplay of factors, with central sensitization playing a pivotal role. This process, characterized by heightened neuronal excitability within the central nervous system, amplifies pain signals and can lead to persistent pain even after the initial injury has healed. Therefore, a crucial aspect of CPSP prevention lies in disrupting the afferent nociceptive signals transmitted from the injured tissues to the spinal cord and brain, thereby preventing the establishment and perpetuation of central sensitization.

While opioids have traditionally been the mainstay of postoperative pain management, their use is not without significant drawbacks. Opioids can have dose-dependent side effects, including respiratory depression, nausea, and constipation. Furthermore, prolonged opioid use can lead to tolerance, opioid-induced hyperalgesia, and an increased risk of chronic opioid use. Recognizing these limitations, the current emphasis in pain management is on multimodal analgesia strategies that incorporate non-opioid medications and regional anaesthesia techniques to optimize pain control while minimizing the risks associated with opioid use.

Non-steroidal anti-inflammatory drugs (NSAIDs) offer a valuable adjunct in pain management, but their use in cardiac surgery is often limited due to concerns regarding bleeding complications and potential renal impairment. Other non-opioid analgesics, such as paracetamol and gabapentinoids, have shown limited efficacy in managing the intense pain associated with sternotomy. Regional anaesthesia techniques have emerged as promising strategies for both acute pain management and potential CPSP prevention in various surgical settings. Techniques such as epidural anaesthesia and paravertebral blocks have demonstrated efficacy in reducing postoperative pain intensity and opioid requirements. However, their application in cardiac surgery presents unique challenges. Epidural anaesthesia carries the risk of neuraxial hematoma due to systemic anticoagulation and heparinization, while paravertebral blocks may be associated with complications such as pneumothorax and pleural puncture. Erector spinae plane block (ESPB) has shown inconsistent results in reducing postoperative pain and morphine consumption in cardiac surgery. Parasternal plane blocks offer advantages over neuraxial techniques but may not adequately address visceral pain.

While regional anaesthesia is crucial for managing acute postoperative pain, its impact on CPSP remains largely unknown. The potential for regional anaesthesia to reduce CPSP has been identified as one of the top research priorities in anaesthesia and perioperative care. Intertransverse process block (ITPB) is a novel and promising alternative, targeting the paravertebral space through extra- paravertebral injection within the intertransverse tissue complex, posterior to the superior costotransverse ligament (SCTL). Recent MRI studies have demonstrated consistent spread of local anaesthetic to the ipsilateral intercostal, paravertebral spaces, neural foramina, and epidural space following ITPB, suggesting potential for both somatic and visceral analgesia. It demonstrated preferential spread of LA to the epidural space and neural foramina over the ESPB, and into the thoracic paravertebral space with effective analgesia after breast and video-assisted thoracoscopic surgeries. Compared to other regional techniques in cardiac surgery, ITPB may offer a simpler and safer approach with reduced risk of pleural puncture and bleeding. Therefore, this trial will assess the efficacy of ITPB in quality of recovery after cardiac surgery, and the potential to mitigate both acute and chronic postsurgical pain in cardiac surgical patients.

Study Design:

Single-centre, prospective, randomized, placebo-controlled, double-blinded trial

Randomization and Concealment Randomisation will be performed in 1:1 ratio using the REDCap randomisation module in the study database, allocating participants to either the ITPB (intervention) or control group in randomly permuted blocks of size four. Sequentially numbered, coded, sealed, opaque envelopes, each containing the group assignment of either interventional or control are then prepared by a third party who takes no further part in the study. The ITPB syringes will be prepared under strict aseptic conditions by a nurse not involved in the study, with blind labelling. The surgical team, blinded to group allocation, will perform standardised surgical procedures. Anaesthetists and nurses responsible for data collection in both ICU and wards are also blinded to the treatment allocation.

Anaesthesia and Interventions All patients receive standard cardiac surgery monitoring. General anaesthesia is induced with midazolam 0.01-0.05 mg/kg, fentanyl 2-5 mcg/kg, and rocuronium 0.5-1 mg/kg to facilitate intubation. Anaesthesia is maintained with sevoflurane and propofol infusion, targeting a Bispectral Index of 40-60. ITPB is performed after anaesthesia induction with the patient in lateral decubitus positioning. Intraoperative opioids (fentanyl and morphine) will be administered at the discretion of the anaesthesiologist. The postoperative analgesia protocol was identical in both study groups, including patient-controlled analgesia (PCA) morphine protocol for 72 hours after surgery, oral analgesics (paracetamol 1g every 6 hours, dihydrocodeine 30mg three times a day), and on-demand antiemetics (intravenous ondansetron 4mg every 8 hours). Rescue analgesics on top of the protocol regimen can be prescribed as needed. Upon ICU admission, propofol infusion is stopped to facilitate weaning from ventilator using Adaptive Support Ventilation (ASV), which adjusts the ventilation parameters depending on the patent's lung mechanics and effort. Pain will be assessed regularly in ICU and on the ward. Upon extubation, pain scores are assessed at 2-hour, 4-hour, 8-hour, 12-hour, 24-hour, 48-hour and 72-hour. Patients receive PCA morphine for moderate to severe pain. Nausea, vomiting and rescue antiemetics are documented.

Ultrasound Block Placement The intervention group received bilateral ITPB after GA induction, whilst sham blocks are performed in the control group. All blocks are performed by an anaesthesiologist who had previously performed ≥50 successful ITPB blocks, using Philips EPIQ ultrasound system, with a curved array transducer (C5-1), and 80mm echogenic nerve block needle (SonoTAP; PAJUNK, Germany). ITPB is performed with the patients positioned in a lateral decubitus position. The target intervertebral level (T4-5) is identified and marked in the preview ultrasound scan. The transducer is placed 2-3 cm lateral to the spinous process. Under strict asepsis, a single-level (T4-5) ultrasound-guided ITPB is performed with the in-plane insertion of the block needle from lateral to medial direction until its tip is at the medial aspect of the retro-SCTL space. After confirming the needle position by distension of the retro-SCTL space after a test bolus injection of 1-2 ml 0.9% normal saline, 20 ml 0.25% levobupivacaine or placebo is injected via the nerve block needle in small aliquots. The same procedure is repeated on the other side with the same volume of study medication. The time required to perform the block will be recorded as the time from insertion of block needle to removal from the patient after injection.

Data Collection All data is collected by research team members blinded to group assignment. Patient demographics and body mass index are recorded. Cumulated opioid consumption data and time to first morphine rescue are extracted from PCA pump. At 2-hour, 4-hour, 8-hour, 12-hour, 24-hour, 48-hour and 72-hour post-extubation, pain scores at rest and on coughing are quantified using NRS from 0 to 10. Zero represents no pain at all while 10 points represents the worst pain ever. The patients are asked to rate the overall satisfaction to pain management on a verbal analogue scale (0=worst possible, 100=best possible) at the predefined points. Any nausea and vomiting, and use of rescue antiemetics are documented. The Chinese validated QoR-15 will be completed at baseline (preoperatively) and postoperatively at 24-hour and 72-hour after extubation. The SF-MPQ- 2 and BPI will be used to evaluate the CPSP at 3-month, 6-month and 12-month after surgery.

Statistics and sample size calculation Sample size was calculated using G*Power software version 3.1.9.3 (Kiel University, Kiel, Germany), based on the QoR-15 score at 24 hours postoperatively the primary outcome. The minimum clinically important difference (MCID) for the QoR-15 score is eight points, and the typical standard deviation (SD) ranges from 10 to 16. Assuming a two-sided type I error of 0.05, type II error of 0.2, and a population variance of 144 (SD = 12), a sample size of 36 per group is required. Allowing for a 20% dropout rate, a total of 96 patients (48 patients per group) will provide 80% power to detect a mean difference of ≥8 points in the QoR-15 score at 24 hours between the two groups.

All outcomes will be analysed and reported on an intention-to-treat basis, with patients analysed according to their randomised group regardless of protocol adherence. A secondary per protocol analysis will be conducted for patients who do not adhere fully to the study protocol. Given the repeated measures of pain scores over time, which are correlated, Generalised Estimating Equation (GEE) models will be used to assess the time effects of postoperative analgesia. Categorical data will be reported as counts and percentages. Continuous variables will be presented as mean (standard deviation) or median (interquartile range), depending on normality assessed using the Shapiro-Wilk's test. Between-group comparison will be conducted using the independent sample t-test for parametric data and Mann-Whitney U test for nonparametric data. Categorical variables will be compared using the Chi-square test. Data analyses will be performed using SPSS 27.0 (IBM Corp, Armonk, NY), and GEE modelling will be conducted using Stata V.14 (Statam College Station, Texas, USA), with a Gaussian distribution, identify-link function, exchangeable correlation structure, and robust standard errors. A P-value of <0.05 will be considered statistically significant, without adjusting for multiple comparisons.

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged 18 or older
* undergoing elective CABG, valve repair/replacement, or combined CABG/valve procedure via sternotomy

Exclusion Criteria:

* Emergency surgery
* redo surgery
* history of chronic pain or being on chronic opioids/sedatives
* renal failure with an estimated glomerular filtration rate ≤30 ml/min (calculated by Cockcroft-Gault formula)
* re-operation within 24 hours after surgery
* intraoperative use of remifentanil
* inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Quality of recovery at 24 hours after extubation | 24 hours after extubation
  The score ranges from 0 to 150, with higher scores associated with better quality of recovery. Though acute pain is identified as an important predictor for the development of CPSP, advanced pain management strategies have failed to reduce the overall incidence of CPSP, suggesting a complex underlying mechanism. Evidence have demonstrated that pain-related functional interference and patient-reported outcomes, such as quality of recovery, might be associated with the development of CPSP. Thus, the primary outcome of this study is the Quality of Recovery (QoR-15) score at 24 hours after extubation. QoR is recommended for patient's comfort after surgery, and is highly valid and reliable patient-centred outcome measure.

SECONDARY OUTCOMES:
Numerical rating scale | 2-hour, 4-hour, 8-hour, 12-hour, 24-hour, 48-hour and 72-hour after extubation
  Pain scores after extubation. It is a 11-points scale from 0 to 10, with zero score means no pain, and 10 score means the worst pain ever
Patient satisfaction with pain management | 2-hour, 4-hour, 8-hour, 12-hour, 24-hour, 48-hour and 72-hour after extubation
  Assessment on patient satisfaction with pain management at predefined time point after extubation. The patients are asked to rate the overall satisfaction to pain management on a verbal analogue scale (0=worst possible, 100=best possible)
Postoperative morphine consumption | 2-hour, 4-hour, 8-hour, 12-hour, 24-hour, 48-hour and 72-hour after extubation
  Postoperative morphine consumption at predefined time point after extubation
Time for first morphine rescue | Up to postoperative day 3, with time of first morphine required recorded
  Time for first morphine rescue (in minutes)
Intraoperative opioid consumption | Intraoperative record
  Converted into morphine equivalence
Duration of mechanical ventilation | Up to postoperative day 1, ventilation requirement will be observed with duration of ventilation required after operation recorded.
  Duration of mechanical ventilation required in postoperative period
Length of stay in ICU and hospital | Up to 1 month after surgery, length of stay in intensive care unit and hospital will be recorded
  Length of ICU and hospital stay postoperatively
Number of episodes of postoperative nausea and vomiting | Perioperative up to 7 days
  Side effects associated with opioids such as postoperative nausea and vomiting (PONV)
Percentage and number of patients having chronic post-surgical pain | 3 month, 6 month and 12 month after surgery
  Incidence of chronic post-surgical pain, which will be asked based on the definition of chronic post-surgical pain by International Association for Study of Pain (IASP)
Pain interference with SF-MPQ-2 | 3 month after surgery
  Together 22-items, each item ranges from 0 to 10. The higher the score, the worst the outcome. Pain interference measured with Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2)
Pain interference with SF-MPQ-2 | 6 month after surgery
  Together 22-items, each item ranges from 0 to 10. The higher the score, the worst the outcome. Pain interference measured with Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2)
Pain interference with SF-MPQ-2 | 12 month after surgery
  Together 22-items, each item ranges from 0 to 10. The higher the score, the worst the outcome. Pain interference measured with Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2)
Pain interference with BPI | 3 month after surgery
  11-items, each item ranges from 0 to 10. The higher the score, the worst the outcome. Pain interference measured with Brief Pain Inventory (BPI) Interference Scale
Pain interference with BPI | 6 month after surgery
  11-items, each item ranges from 0 to 10. The higher the score, the worst the outcome. Pain interference measured with Brief Pain Inventory (BPI) Interference Scale
Pain interference with BPI | 12 month after surgery
  11-items, each item ranges from 0 to 10. The higher the score, the worst the outcome. Pain interference measured with Brief Pain Inventory (BPI) Interference Scale
Number of episodes requested antiemetics after surgery | Up to postoperative day 7
  The number of times the patient requesting antiemetic for nausea and vomiting will be documented

CONTACTS AND LOCATIONS:
Overall Officials: Henry Wong, Principal Investigator — Hospital Authority

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhang H, Qu Z, Miao Y, Zhang Y, Qian L, Hua B, Hua Z. Comparison between ultrasound-guided multi-injection intertransverse process and thoracic paravertebral blocks for major breast cancer surgery: a randomized non-inferiority trial. Reg Anesth Pain Med. 2023 Apr;48(4):161-166. doi: 10.1136/rapm-2022-104003. Epub 2022 Dec 15. PMID 36522043
- [Result] Moorthy A, Ni Eochagain A, Dempsey E, Wall V, Marsh H, Murphy T, Fitzmaurice GJ, Naughton RA, Buggy DJ. Postoperative recovery with continuous erector spinae plane block or video-assisted paravertebral block after minimally invasive thoracic surgery: a prospective, randomised controlled trial. Br J Anaesth. 2023 Jan;130(1):e137-e147. doi: 10.1016/j.bja.2022.07.051. Epub 2022 Sep 13. PMID 36109206
- [Result] Myles PS, Myles DB, Galagher W, Chew C, MacDonald N, Dennis A. Minimal Clinically Important Difference for Three Quality of Recovery Scales. Anesthesiology. 2016 Jul;125(1):39-45. doi: 10.1097/ALN.0000000000001158. PMID 27159009
- [Result] Bu XS, Zhang J, Zuo YX. Validation of the Chinese Version of the Quality of Recovery-15 Score and Its Comparison with the Post-Operative Quality Recovery Scale. Patient. 2016 Jun;9(3):251-9. doi: 10.1007/s40271-015-0148-6. PMID 26518201
- [Result] Ger LP, Ho ST, Sun WZ, Wang MS, Cleeland CS. Validation of the Brief Pain Inventory in a Taiwanese population. J Pain Symptom Manage. 1999 Nov;18(5):316-22. doi: 10.1016/s0885-3924(99)00087-1. PMID 10584454
- [Result] Tsui FPY, Wong SSC, Chan TCW, Lee Y, Cheung CW. A validation study of the Cantonese Chinese version of short form McGill pain questionnaire 2 in Cantonese-speaking patients with chronic pain in Hong Kong. Pain Pract. 2024 Mar;24(3):449-457. doi: 10.1111/papr.13319. Epub 2023 Nov 17. PMID 37975327
- [Result] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725
- [Result] Maurice-Szamburski A, Bringuier S, Auquier P, Capdevila X. From pain level to pain experience: redefining acute pain assessment to enhance understanding of chronic postsurgical pain. Br J Anaesth. 2024 Nov;133(5):1021-1027. doi: 10.1016/j.bja.2024.08.003. Epub 2024 Sep 26. PMID 39332996
- [Result] Karmakar MK, Sivakumar RK, Sheah K, Pangthipampai P, Lonnqvist PA. The Retro Superior Costotransverse Ligament Space as a New Target for Ultrasound-Guided Intertransverse Process Block: A Report of 2 Cases. A A Pract. 2022 Jul 22;16(7):e01610. doi: 10.1213/XAA.0000000000001610. eCollection 2022 Jul 1. PMID 35867848
- [Result] Bhoi D, Narasimhan P, Nethaji R, Talawar P. Ultrasound-Guided Midpoint Transverse Process to Pleura Block in Breast Cancer Surgery: A Case Report. A A Pract. 2019 Feb 1;12(3):73-76. doi: 10.1213/XAA.0000000000000850. PMID 30085935
- [Result] Pangthipampai P, Siriwanarangsun P, Pakpirom J, Sivakumar RK, Karmakar MK. Intertransverse process block (ITPB) at the retro-superior costotransverse ligament (retro-SCTL) space: Evaluation of local anesthetic spread using MRI and sensory blockade in healthy volunteers. J Clin Anesth. 2025 Feb;101:111718. doi: 10.1016/j.jclinane.2024.111718. Epub 2024 Dec 18. PMID 39700657
- [Result] Costache I, de Neumann L, Ramnanan CJ, Goodwin SL, Pawa A, Abdallah FW, McCartney CJL. The mid-point transverse process to pleura (MTP) block: a new end-point for thoracic paravertebral block. Anaesthesia. 2017 Oct;72(10):1230-1236. doi: 10.1111/anae.14004. Epub 2017 Aug 1. PMID 28762464
- [Result] Bowness JS, Pawa A, Turbitt L, Bellew B, Bedforth N, Burckett-St Laurent D, Delbos A, Elkassabany N, Ferry J, Fox B, French JLH, Grant C, Gupta A, Harrop-Griffiths W, Haslam N, Higham H, Hogg R, Johnston DF, Kearns RJ, Kopp S, Lobo C, McKinlay S, Memtsoudis S, Merjavy P, Moka E, Narayanan M, Narouze S, Noble JA, Phillips D, Rosenblatt M, Sadler A, Sebastian MP, Taylor A, Thottungal A, Valdes-Vilches LF, Volk T, West S, Wolmarans M, Womack J, Macfarlane AJR. International consensus on anatomical structures to identify on ultrasound for the performance of basic blocks in ultrasound-guided regional anesthesia. Reg Anesth Pain Med. 2022 Feb;47(2):106-112. doi: 10.1136/rapm-2021-103004. Epub 2021 Sep 22. PMID 34552005
- [Result] Lewis O, Lloyd J, Ferry J, Macfarlane AJR, Womack J, El-Boghdadly K, Shelton CL, Schaff O, Quick TJ, Smith AF, Cannons K, Pearson A, Heelas L, Rodger D, Marshall J, Pellowe C, Bowness JS, Kearns RJ. Regional anaesthesia research priorities: a Regional Anaesthesia UK (RA-UK) priority setting partnership involving patients, carers and healthcare professionals. Anaesthesia. 2025 Feb;80(2):170-178. doi: 10.1111/anae.16473. Epub 2024 Nov 25. PMID 39584463
- [Result] Capuano P, Sepolvere G, Toscano A, Scimia P, Silvetti S, Tedesco M, Gentili L, Martucci G, Burgio G. Fascial plane blocks for cardiothoracic surgery: a narrative review. J Anesth Analg Crit Care. 2024 Mar 11;4(1):20. doi: 10.1186/s44158-024-00155-5. PMID 38468350
- [Result] Wong HMK, Chen PY, Tang GCC, Chiu SLC, Mok LYH, Au SSW, Wong RHL. Deep Parasternal Intercostal Plane Block for Intraoperative Pain Control in Cardiac Surgical Patients for Sternotomy: A Prospective Randomized Controlled Trial. J Cardiothorac Vasc Anesth. 2024 Mar;38(3):683-690. doi: 10.1053/j.jvca.2023.11.038. Epub 2023 Nov 30. PMID 38148266
- [Result] Sorenstua M, Zantalis N, Raeder J, Vamnes JS, Leonardsen AL. Spread of local anesthetics after erector spinae plane block: an MRI study in healthy volunteers. Reg Anesth Pain Med. 2023 Feb;48(2):74-79. doi: 10.1136/rapm-2022-104012. Epub 2022 Nov 9. PMID 36351741
- [Result] Oostvogels L, Weibel S, Meissner M, Kranke P, Meyer-Friessem CH, Pogatzki-Zahn E, Schnabel A. Erector spinae plane block for postoperative pain. Cochrane Database Syst Rev. 2024 Feb 12;2(2):CD013763. doi: 10.1002/14651858.CD013763.pub3. PMID 38345071
- [Result] Karmakar MK, Lonnqvist PA. The clinical use of the thoracic erector spinae plane block. Con - ESPB is not useful for thoracic analgesia. J Clin Anesth. 2024 May;93:111353. doi: 10.1016/j.jclinane.2023.111353. Epub 2023 Nov 30. No abstract available. PMID 38039630
- [Result] Dost B, De Cassai A, Balzani E, Tulgar S, Ahiskalioglu A. Effects of ultrasound-guided regional anesthesia in cardiac surgery: a systematic review and network meta-analysis. BMC Anesthesiol. 2022 Dec 29;22(1):409. doi: 10.1186/s12871-022-01952-7. PMID 36581838
- [Result] Macaire P, Ho N, Nguyen T, Nguyen B, Vu V, Quach C, Roques V, Capdevila X. Ultrasound-Guided Continuous Thoracic Erector Spinae Plane Block Within an Enhanced Recovery Program Is Associated with Decreased Opioid Consumption and Improved Patient Postoperative Rehabilitation After Open Cardiac Surgery-A Patient-Matched, Controlled Before-and-After Study. J Cardiothorac Vasc Anesth. 2019 Jun;33(6):1659-1667. doi: 10.1053/j.jvca.2018.11.021. Epub 2018 Nov 19. PMID 30665850
- [Result] Wang W, Yang W, Liu A, Liu J, Yuan C. The Analgesic Effect of Ultrasound-guided Erector Spinae Plane Block in Median Sternotomy Cardiac Surgery in Adults: A Systematic Review and Meta-analysis of Randomized Controlled Trials. J Cardiothorac Vasc Anesth. 2024 Nov;38(11):2792-2800. doi: 10.1053/j.jvca.2024.05.019. Epub 2024 May 22. PMID 38890084
- [Result] Richardson J, Lonnqvist PA, Naja Z. Bilateral thoracic paravertebral block: potential and practice. Br J Anaesth. 2011 Feb;106(2):164-71. doi: 10.1093/bja/aeq378. PMID 21233114
- [Result] Kukreja, P., Paul, L.M., Sellers, A.R. The Role of Regional Anesthesia in the Development of Chronic Pain: a Review of Literature. Curr Anesthesiol Rep 12, 417 - 438 (2022). https://doi.org/10.1007/s40140-022-00536-y
- [Result] Andreae MH, Andreae DA. Regional anaesthesia to prevent chronic pain after surgery: a Cochrane systematic review and meta-analysis. Br J Anaesth. 2013 Nov;111(5):711-20. doi: 10.1093/bja/aet213. Epub 2013 Jun 28. PMID 23811426
- [Result] Naganuma M, Tokita T, Sato Y, Kasai T, Kudo Y, Suzuki N, Masuda S, Nagaya K. Efficacy of Preoperative Bilateral Thoracic Paravertebral Block in Cardiac Surgery Requiring Full Heparinization: A Propensity-Matched Study. J Cardiothorac Vasc Anesth. 2022 Feb;36(2):477-482. doi: 10.1053/j.jvca.2021.05.001. Epub 2021 May 13. PMID 34099376
- [Result] Zhou K, Li D, Song G. Comparison of regional anesthetic techniques for postoperative analgesia after adult cardiac surgery: bayesian network meta-analysis. Front Cardiovasc Med. 2023 May 22;10:1078756. doi: 10.3389/fcvm.2023.1078756. eCollection 2023. PMID 37283577
- [Result] Verret M, Lauzier F, Zarychanski R, Perron C, Savard X, Pinard AM, Leblanc G, Cossi MJ, Neveu X, Turgeon AF; Canadian Perioperative Anesthesia Clinical Trials (PACT) Group. Perioperative Use of Gabapentinoids for the Management of Postoperative Acute Pain: A Systematic Review and Meta-analysis. Anesthesiology. 2020 Aug;133(2):265-279. doi: 10.1097/ALN.0000000000003428. PMID 32667154
- [Result] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Result] Hah JM, Bateman BT, Ratliff J, Curtin C, Sun E. Chronic Opioid Use After Surgery: Implications for Perioperative Management in the Face of the Opioid Epidemic. Anesth Analg. 2017 Nov;125(5):1733-1740. doi: 10.1213/ANE.0000000000002458. PMID 29049117
- [Result] Gutwinski S, Schoofs N, Stuke H, Riemer TG, Wiers CE, Bermpohl F. Opioid tolerance in methadone maintenance treatment: comparison of methadone and levomethadone in long-term treatment. Harm Reduct J. 2016 Feb 16;13:7. doi: 10.1186/s12954-016-0095-0. PMID 26879120
- [Result] Choiniere M, Watt-Watson J, Victor JC, Baskett RJ, Bussieres JS, Carrier M, Cogan J, Costello J, Feindel C, Guertin MC, Racine M, Taillefer MC. Prevalence of and risk factors for persistent postoperative nonanginal pain after cardiac surgery: a 2-year prospective multicentre study. CMAJ. 2014 Apr 15;186(7):E213-23. doi: 10.1503/cmaj.131012. Epub 2014 Feb 24. PMID 24566643
- [Result] Gjeilo KH, Stenseth R, Wahba A, Lydersen S, Klepstad P. Chronic postsurgical pain in patients 5 years after cardiac surgery: A prospective cohort study. Eur J Pain. 2017 Mar;21(3):425-433. doi: 10.1002/ejp.918. Epub 2016 Jul 26. PMID 27461370
- [Result] Meyerson J, Thelin S, Gordh T, Karlsten R. The incidence of chronic post-sternotomy pain after cardiac surgery--a prospective study. Acta Anaesthesiol Scand. 2001 Sep;45(8):940-4. doi: 10.1034/j.1399-6576.2001.450804.x. PMID 11576043
- [Result] Kalso E, Mennander S, Tasmuth T, Nilsson E. Chronic post-sternotomy pain. Acta Anaesthesiol Scand. 2001 Sep;45(8):935-9. doi: 10.1034/j.1399-6576.2001.450803.x. PMID 11576042
- [Result] Eisenberg E, Pultorak Y, Pud D, Bar-El Y. Prevalence and characteristics of post coronary artery bypass graft surgery pain (PCP). Pain. 2001 May;92(1-2):11-7. doi: 10.1016/s0304-3959(00)00466-8. PMID 11323122
- [Result] Sandkuhler J, Gruber-Schoffnegger D. Hyperalgesia by synaptic long-term potentiation (LTP): an update. Curr Opin Pharmacol. 2012 Feb;12(1):18-27. doi: 10.1016/j.coph.2011.10.018. Epub 2011 Nov 9. PMID 22078436
- [Result] Woolf CJ, Chong MS. Preemptive analgesia--treating postoperative pain by preventing the establishment of central sensitization. Anesth Analg. 1993 Aug;77(2):362-79. doi: 10.1213/00000539-199377020-00026. No abstract available. PMID 8346839
- [Result] Ong CK, Lirk P, Seymour RA, Jenkins BJ. The efficacy of preemptive analgesia for acute postoperative pain management: a meta-analysis. Anesth Analg. 2005 Mar;100(3):757-773. doi: 10.1213/01.ANE.0000144428.98767.0E. PMID 15728066
- [Result] Katz J, Clarke H, Seltzer Z. Review article: Preventive analgesia: quo vadimus? Anesth Analg. 2011 Nov;113(5):1242-53. doi: 10.1213/ANE.0b013e31822c9a59. Epub 2011 Sep 30. PMID 21965352
- [Derived] Wong HMK, Sivakumar RK, Wong WT, Chan AKM, Yeung ZHS, Chen PY, Tang STW, Chu MHM, Wong RHL, Ho KM. Intertransverse process block to improve quality of recovery and pain management in cardiac surgery: Protocol for a double-blinded randomized controlled trial. PLoS One. 2025 Sep 24;20(9):e0328954. doi: 10.1371/journal.pone.0328954. eCollection 2025. PMID 40991544